CLINICAL TRIAL: NCT02040194
Title: Efficacy and Safety of AM-101 in the Treatment of Acute Peripheral Tinnitus 3
Brief Title: AM-101 in the Treatment of Acute Tinnitus 3
Acronym: TACTT3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Auris Medical AG (Industry)
Responsible Party: Sponsor
Organization: Auris Medical, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AM-101-CL-12-02
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — PDCD5 protein, rat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AM-101 injection (Experimental): AM-101
  Interventions: Drug: AM-101
- Placebo injection (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AM-101 — AM-101 gel for intratympanic injection
  Arms: AM-101 injection
Drug: Placebo — Placebo gel for intratympanic injection
  Arms: Placebo injection

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of the study drug, AM-101. AM-101 is tested for the treatment of tinnitus that started as the result of an injury to the inner ear or due to middle ear inflammation (otitis media). Subjects with tinnitus can take part in the study, if their tinnitus started within the last 3 months or within the last >3 to 6 months.

DETAILED DESCRIPTION:
This phase III study is assessing the drug's safety and is aiming to demonstrate efficacy of repeated intratympanic AM-101 injections in the treatment of acute peripheral tinnitus (up to 3 months (Stratum A), or between >3 and 6 months (Stratum B) from onset).

ELIGIBILITY:
Inclusion Criteria:

1. Persistent subjective peripheral tinnitus (unilateral or bilateral) following traumatic cochlear injury (acute acoustic trauma, blast trauma, middle ear surgery, inner ear barotrauma, tympanic membrane trauma) or otitis media with onset no longer than 3 months (Stratum A) or between >3 months and 6 months (Stratum B) prior to randomization, as documented by medical report or by documented medical history. Upon implementation of protocol amendment 6, subjects with tinnitus following traumatic cochlear injury will only be eligible if they are affected only unilaterally.
2. Age ≥ 18 years and ≤ 75 years;
3. Negative pregnancy test (woman of childbearing potential);
4. Willing and able to use adequate hearing protection, respectively to refrain from engaging in activities or work involving loud noise exposure where sufficient hearing protection is not possible or ensured;
5. Willing and able to protect ear canal and middle ear from water exposure as long as tympanic membrane is not fully closed.

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

1. Fluctuating tinnitus;
2. Intermittent tinnitus;
3. Tinnitus resulting from traumatic head or neck injury;
4. Presence of chronic tinnitus;
5. Meniere's Disease, history of endolymphatic hydrops, or history of fluctuating hearing loss;
6. History of repeated idiopathic sudden sensorineural hearing loss or history of acoustic neuroma;
7. Ongoing acute or chronic otitis media or otitis externa;
8. Other treatment of tinnitus for the study duration;
9. Known hypersensitivity, allergy or intolerance to the study medication or any history of severe, abnormal drug reaction;
10. Women who are breast-feeding, pregnant or who are planning to become pregnant during the study;
11. Women of childbearing potential who are unwilling or unable to practice contraception, such as hormonal contraceptives, double barrier, sexual abstinence or intercourse with a partner who has been vasectomised for at least three months;
12. Concurrent participation in another clinical study or participation in another clinical study within 30 days prior to randomization.

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 893 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint - alternate primary efficacy endpoints: Tinnitus Functional Index (TFI) | Baseline to Day 84
  Improvement in TFI total score
Efficacy endpoint - alternate primary efficacy endpoints: Patient-reported Tinnitus loudness on a Numerical Rating Scale (TLQ NRS loudest) | Baseline to Day 84
  Improvement in TLQ NRS loudest
Safety endpoint: Hearing threshold | Baseline to Day 35
  Occurrence of deterioration in hearing threshold >= 15 decibel (dB) at the average of two contiguous test frequencies (air conduction) in the treated ear(s)

SECONDARY OUTCOMES:
Efficacy endpoint - TFI | Baseline to Day 10 and Day 35
  Improvement in TFI total score
Efficacy endpoint - TLQ NRS loudest | Baseline to Day 10 and Day 35
  Improvement in patient-reported tinnitus loudness
Efficacy endpoint - patient-reported tinnitus annoyance (TAQ NRS worst) | Baseline to Day10, Day 35 and Day 84
  Improvement in TAQ NRS worst
Efficacy endpoint - TFI sleep score | Baseline to Day10, Day 35 and Day 84
  Improvement in TFI sleep score. The subscale "sleep" will be evaluated only for subjects with a TFI Sleep score greater than 0 at baseline.
Efficacy endpoint - Patient global impression of change in tinnitus severity (PGIC Tinnitus) | at Day10, Day 35 and Day 84
  Patient global impression of change in tinnitus severity
Safety endpoint - Hearing threshold | Baseline to Day 1, Day 2, Day 10 and Day 84
  Occurrence of deterioration in hearing threshold >= 15 dB at the average of two contiguous test frequencies in the treated ear(s)
Safety endpoint - Hearing threshold | Baseline to Day 1, Day 2, Day 10 and Day 84
  Difference in occurrence of deterioration in hearing threshold >= 15 dB at the average of two contiguous test frequencies between the treated and untreated contralateral ear (subjects with unilaterally treated tinnitus only)
Safety endpoint - AEs and SAEs | Up to Day 84
  Occurence and severity of adverse events (AEs) and serious adverse Events (SAEs), differentiated by relatedness, and by treatment-emergence and procedure-emergence

CONTACTS AND LOCATIONS:
Locations (1):
- Please check the study webpage below for a study site list, Munich, Germany

REFERENCES:
- See also: Link to Result entry in clinicaltrialsregister.eu — https://www.clinicaltrialsregister.eu/ctr-search/trial/2012-004099-20/results